CLINICAL TRIAL: NCT06965257
Title: Continuous Non-invasive Blood Pressure Monitoring During Carotid Endarterectomy Surgery
Brief Title: Non-invasive Blood Pressure Monitoring in Carotid Surgery
Acronym: SPARK
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250362; 2025-A00444-45 (Other: ID RCB)
Record Dates: First submitted 2025-04-14; First posted 2025-05-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Carotid Endarterectomy Surgery
Keywords: Prospective study; Non-invasive blood pressure monitoring; Carotid endarterectomy surgery; Anaesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Continuous non-invasive blood pressure monitoring — Addition prior to anaesthetic induction of the non-invasive monitoring device (digital sleeve available at the investigation site) for blood pressure measurement on the side ipsilateral to the arterial catheter

SUMMARY:
Carotid endarterectomy surgery carries significant neurological and cardiac risks, requiring continuous monitoring of blood pressure. In standard practice, this monitoring is carried out using an arterial catheter inserted at the start of the operation. This invasive procedure is generally not well received by the patient and is a source of potential ischaemic and infectious complications.

The use of a non-invasive extracorporeal device (digital cuff) for continuous measurement of arterial pressure, based on detection of the pulse wave by plethysmography, could provide an interesting alternative. Nevertheless, the concordance of blood pressure curves measured continuously by the arterial catheter and by non-invasive pulse wave analysis remains insufficiently studied for carotid endarterectomy surgery.

The aim of this study was to evaluate the concordance, using the Bland-Altman method, of mean arterial pressure curves measured continuously by the invasive arterial catheter (standard management) and by non-invasive pulse wave contour analysis (non-invasive extracorporeal sensor) in carotid endarterectomy surgery.

This was a non-interventional study. Patient management is carried out according to current recommendations for carotid endarterectomy surgery: placement of an arterial catheter at the start of the procedure and frontal NIRS electrodes.

A non-invasive monitoring device (ClearSight™ digital cuff available on the investigation site) will then be added to measure blood pressure on the side ipsilateral to the arterial catheter.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients undergoing carotid endarterectomy surgery under general anesthetic
* Patient who has been informed and has not objected

Exclusion Criteria:

* Technical or physical impossibility of inserting an arterial catheter or extracorporeal sensor (digital cuff)
* Patient of legal age unable to express his/her opposition
* Patient under guardianship, curatorship or legal protection
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing carotid endarterectomy under general anaesthesia
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Bland-Altman concordance analysis (accuracy, reproducibility and limits of agreement) between mean arterial pressures measured invasively (arterial catheter) and non-invasively (extracorporeal sensor) | through operative care procedure, [beginning of procedure ; end of procedure]
  Concordance between mean arterial pressures measured by the invasive arterial catheter (standard management) and by a non-invasive extracorporeal sensor (study method) during the different phases of the care procedure

SECONDARY OUTCOMES:
Bland-Altman concordance analyses (accuracy, reproducibility and limits of agreement) between systolic and diastolic arterial pressures measured invasively (arterial catheter) and non-invasively (extracorporeal sensor) | through operative care procedure, [beginning of procedure ; end of procedure]
  Measurement concordance for systolic and diastolic blood pressures
Focus on the successive phases of the procedure: anaesthetic induction, before, during and after carotid clamping | through operative care procedure, [beginning of procedure ; end of procedure]
  Concordance of measurements during the different phases of surgery (anaesthetic induction then before, during and after carotid clamping)
Invasive arterial pressure (measured in mmHg) | through operative care procedure, [beginning of procedure ; end of procedure]
  Relationship between invasive arterial pressure (measured in mmHg) and clinical parameters using regression model type y = f(x).
Non-invasive arterial pressure (measured in mmHg) | through operative care procedure, [beginning of procedure ; end of procedure]
  Relationship between non-invasive arterial pressure (measured in mmHg) and clinical parameters using regression model type y = f(x).
NIRS (measured in %) | through operative care procedure, [beginning of procedure ; end of procedure]
  Relationship between NIRS (measured in %) and clinical parameters using regression model type y = f(x).
Search for measurement bias according to operators using regression models | through operative care procedure, [beginning of procedure ; end of procedure]
  Identify any confounding variables (arrhythmias, operators)

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU Henri Mondor - DMU CARE, Créteil, France, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION